CLINICAL TRIAL: NCT03711370
Title: A Pilot-Feasibility of a Home-based Intervention to Reduce Obesity Risk for Bottle-fed Infants
Brief Title: Opaque Bottle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Ventura, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-164-CP; R21HD096236 (NIH)
Record Dates: First submitted 2018-10-14; First posted 2018-10-18 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Opaque Bottles; Conventional, Clear Bottles
Keywords: infant feeding; feeding interactions; maternal feeding practices; bottle-feeding; opaque bottles
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Intervention Model Description: All participants were randomly assigned to either the opaque bottle group or the clear bottle group. Mothers were asked to use their assigned bottle type to feed their infant for a full 12-week period. Pre-tests were given before the 12-week period and post-tests occured after the 12-week period. During these tests, we observed each mother using the clear bottle to feed her infant on one visit and the opaque bottle on another visit. The order of these conditions was randomized and counterbalanced.
Who Masked: Outcomes Assessor
Masking Description: The video coders were masked during video analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opaque Bottle Group (Experimental): This group was given a set of opaque bottles to use during infant feedings for a full 12-week period.
  Interventions: Other: Opaque Bottle
- Clear Bottle Group (Active Comparator): This group was given a set of clear bottles to use during infant feedings for a full 12-week period.
  Interventions: Other: Clear Bottle

INTERVENTIONS:
Other: Clear Bottle — These mothers received usual care from their pediatric providers and each mother was given 12 conventional, clear bottles of various sizes (4-12 ounces) that were compatible with a variety of different nipples manufactured by leading bottle companies. Mothers were also given handouts about proper formula preparation and paced bottle-feeding, which included messages about feeding in response to infant cues.
  Arms: Clear Bottle Group
Other: Opaque Bottle — These mothers received everything provided to the clear group, but instead received 12 opaque bottles of various sizes (4-12 ounces). These bottles were stainless steel and compatible with a variety of different nipples manufactured by a leading bottle company. Mothers in the intervention group also received an additional handout that contained safety tips for their opaque bottles (e.g., never microwave your bottle).
  Arms: Opaque Bottle Group

SUMMARY:
The proposed research aimed to conduct an intervention study assessing the effect of feeding mode (clear versus opaque bottle) on the quality and outcome of infant feeding interactions.

DETAILED DESCRIPTION:
The overall objective of the proposed pilot/feasibility study was to evaluate a home- and family-based intervention to increase bottle-feeding mothers' responsiveness to infant satiety cues and moderate bottle-feeding infants' rates of weight gain over a 12-week period. Specifically, the investigators propose to provide mothers with opaque, weighted bottles (instead of conventional, clear bottles) with which to feed their infants; based on preliminary studies, it is hypothesized that removal of mothers' abilities to assess the amount the infant consumes during feeding will facilitate abilities to feed in response to infant satiation cues.

For the proposed research, predominantly bottle-feeding mothers with <6-month-old infants were randomized to use opaque bottles (intervention or opaque group) or to use clear bottles (control or clear group). The investigators conducted home-based assessments at the beginning and end of the 12-week study period during which mothers were video-recorded feeding their infants using clear or opaque bottles. Two interim assessments will be conducted (after 2 and 6 weeks) to assess feeding adequacy and fidelity to the intervention. During feeding observations, infant intake were assessed via bottle weight. Video-records were later coded for maternal responsiveness to infant cues using the Nursing Child Assessment Parent-Child Interaction Feeding Scale (NCAFS). It was hypothesized that mothers in the opaque group will feed their infants less and show greater increases in their levels of responsiveness to infant cues compared to mothers in the clear group. Infants' weight and length were measured at the beginning and end of the 12-week study; weight-for-length z-scores (WLZ) were calculated using the World Health Organization (WHO) Growth Standards. It was hypothesized that WLZ change would be significantly lower for infants in the opaque compared to the clear group. The feasibility of the intervention was also explored by collecting and analyzing objective and subjective data related to the extent to which mothers use and like the bottles, and whether characteristics of mothers or infants moderate intervention effects. The proposed feasibility study is a critical step toward understanding mothers' acceptance and use of opaque bottles compared to conventional, clear bottles, and the potential for opaque bottles to improve the outcome of feeding interactions in home-based settings.

ELIGIBILITY:
Inclusion Criteria:

* mothers 18-40-years of age
* infants <24-weeks of age
* predominantly bottle-feeding (>50% of feedings)
* mother predominantly or solely responsible for infant feeding
* dyad has a pediatrician and plans to attend infant well-visits
* mother is willing to use stainless-steel bottles and to provide the study with her current bottles, which would be returned after study completion
* prior to the introduction of solid foods.

Exclusion Criteria:

* preterm birth (i.e., gestational age <37 weeks)
* low birth weight (<2500 g)
* maternal smoking during pregnancy
* current or past medical conditions that interfere with oral feeding
* history of slow growth or failure to thrive
* weight for length percentile <5th
* diagnosed developmental delay (e.g., Down's syndrome)
* currently using opaque bottles

Ages: 0 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- Healthy Kids Laboratory within the French Hospital Copeland Health Education Pavilion, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not currently plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Ventura AK, Pollack Golen R. A pilot study comparing opaque, weighted bottles with conventional, clear bottles for infant feeding. Appetite. 2015 Feb;85:178-84. doi: 10.1016/j.appet.2014.11.028. Epub 2014 Nov 28. PMID 25445988
- [Background] Ventura AK, Hernandez A. Effects of opaque, weighted bottles on maternal sensitivity and infant intake. Matern Child Nutr. 2019 Apr;15(2):e12737. doi: 10.1111/mcn.12737. Epub 2018 Nov 22. PMID 30345622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between December 2018 and May 2022. Mothers with young infants were recruited through local radio station ads; targeted social media ads; Supplemental Nutrition Assistance Program for Women, Infants, and Children (WIC) offices; perinatal education classes; and pediatric offices; as well as through a list of past participants who asked to be notified of future studies.
Pre-assignment Details: Participants engaged in two initial pre-test assessments that occurred in participants' homes or via video conference. Pre-tests were separated by no more than 2 weeks (average time between pre-tests=2.5+/-2.0 days, range=1-8 days). After the second pre-test assessment, participants were randomized to the control or intervention groups.
Groups:
- Clear Bottle Group: This group was given a set of clear bottles that were to be used during infant feedings for a full 12-week period.
  Clear Bottle: These mothers received usual care from their pediatric providers and each mother was given 12 conventional, clear bottles of various sizes (4-12 ounces) that were compatible with a variety of different nipples manufactured by leading bottle companies. Mothers were also given a handouts about proper formula preparation and paced bottle-feeding, which includes messages about feeding in response to infant cues.
- Opaque Bottle Group: This group was given a set of opaque bottles that are to be used during infant feedings for a full 12-week period.
  Opaque Bottle: These mothers received everything provided to the clear group, but instead received 12 opaque, weighted bottles of various sizes (4-12 ounces). These bottles were stainless steel and compatible with a variety of different nipples manufactured by leading bottle companies. Mothers in the intervention group received an additional handout that contained safety tips for their opaque bottles (e.g., never microwave your bottle).
Period: Overall Study
Arm/Group | Clear Bottle Group | Opaque Bottle Group
Started | 76 (38 mother-infant dyads (38 mothers + 38 infants = 76 participants total) were randomized to the Clear Bottle Group) | 76 (38 mother-infant dyads (38 mothers + 38 infants = 76 participants total) were randomized to the Opaque Bottle Group)
Pre-Test: Clear Bottle Feeding Condition | 76 (38 mother-infant dyads (38 mothers + 38 infants = 76 participants total)) | 76 (38 mother-infant dyads (38 mothers + 38 infants = 76 participants total))
Pre-Test: Opaque Bottle Feeding Condition | 76 (38 mother-infant dyads (38 mothers + 38 infants = 76 participants total)) | 76 (38 mother-infant dyads (38 mothers + 38 infants = 76 participants total))
Post-test: Clear Bottle Feeding Condition | 60 (30 mother-infant dyads (30 mothers + 30 infants = 60 participants total)) | 66 (33 mother-infant dyads (33 mothers + 33 infants = 66 participants total))
Post-test: Opaque Bottle Feeding Condition | 60 (30 mother-infant dyads (30 mothers + 30 infants = 60 participants total)) | 66 (33 mother-infant dyads (33 mothers + 33 infants = 66 participants total))
Completed | 60 (30 mother-infant dyads (30 mothers + 30 infants = 60 participants total) in the Clear Bottle Group were included in data analysis) | 60 (30 mother-infant dyads (30 mothers + 30 infants = 60 participants total) in the Opaque Bottle Group were included in data analysis)
Not Completed | 16 | 16
Not completed — Lost to Follow-up | 16 | 10
Not completed — Pre-test or Post-test visits were >2 weeks apart | 0 | 6

BASELINE CHARACTERISTICS:
Population: 38 mother-infant dyads (38 mothers+38 infants=76 participants total) were in the Clear Bottle Group and 38 mother-infant dyads (38 mothers+38 infants=76 participants total) were in the Opaque Bottle Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Bottle Group | Opaque Bottle Group | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] — Mother Age at Study Entry Population: Measure Analysis Population Description: Data are for mothers only (n = 76)
  years
    number analyzed (Participants) | 38 | 38 | 76
    (all) | 31.4 (5.8) | 30.9 (5.2) | 31.1 (5.4)
Age, Continuous [Mean (Standard Deviation); unit: months] — Infant Age at Study Entry Population: Data are for infants only (n = 76)
  months
    number analyzed (Participants) | 38 | 38 | 76
    (all) | 3.0 (1.5) | 2.8 (1.3) | 2.9 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Mothers' sex; self-reported Population: Data are for mothers only (n = 76)
  Participants
    number analyzed (Participants) | 38 | 38 | 76
    Female | 38 | 38 | 76
    Male | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Infant sex; reported by mothers Population: Data are for infants only (n = 76)
  Participants
    number analyzed (Participants) | 38 | 38 | 76
    Female | 25 | 15 | 40
    Male | 13 | 23 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Maternal race/ethnicity was self-reported Population: Data are for mothers only (n = 76)
  Participants
    Race/Ethnicity: number analyzed (Participants) | 38 | 38 | 76
    Race/Ethnicity: Non-Hispanic White | 10 | 8 | 18
    Race/Ethnicity: Hispanic | 26 | 29 | 55
    Race/Ethnicity: Asian | 2 | 0 | 2
    Race/Ethnicity: Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Infant race/ethnicity was reported by mothers Population: Data are for infants only (n = 76)
  Participants
    Race/Ethnicity: number analyzed (Participants) | 38 | 38 | 76
    Race/Ethnicity: Non-Hispanic White | 10 | 8 | 18
    Race/Ethnicity: Hispanic | 26 | 29 | 55
    Race/Ethnicity: Asian | 2 | 0 | 2
    Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 152

OUTCOME MEASURES:

1. Primary Outcome: Infant Intake (mL) During the Observed Feeding
Description: During post-tests, participants in both the Clear Bottle and Opaque Bottle Groups were asked to use the clear bottle during one feeding observation and the opaque bottle during the other feeding across the two post-test assessments, which ensured research assistants remained masked to whether the participant was in the intervention or control group and allowed for within-subject comparison of effects of clear versus opaque bottles on maternal sensitivity and infant intake; order of bottle presentation was counterbalanced.
  For both opaque and clear bottle-feedings, infant intake was assessed by weighing the infant's bottle before and after each feeding observation using a top-loading balance (SP601 Scout Pro Portable Balance, Ohaus, New Jersey, USA).
Time Frame: 12-week period
Population: Overall Number of Participants Analyzed for each group (n=30) is not consistent with the number of participants indicated in the Participant Flow module because data were analyzed at the level of the dyad (n = 30 dyads per group), not at the level of each individual member of the dyad (n = 60 individuals per group, which represents 30 mothers + 30 infants)
Measure: Least Squares Mean (Standard Error); unit: mL
Groups:
- Clear Bottle Group - Clear Bottle Condition; Clear Bottle Group - Opaque Bottle Condition.: The Clear Bottle group was given a set of clear bottles to use during infant feedings for a full 12-week period. These mothers received usual care from their pediatric providers and each mother was given 12 conventional, clear bottles of various sizes (4-12 ounces) that were compatible with a variety of different nipples manufactured by leading bottle companies. Mothers were also given handouts about proper formula preparation and paced bottle-feeding, which included messages about feeding in response to infant cues.
  During post-tests, participants in both the Clear Bottle and Opaque Bottle Groups were asked to use the clear bottle during one feeding observation and the opaque bottle during the other feeding across the two post-test assessments, which ensured research assistants remained masked to whether the participant was in the intervention or control group and allowed for within-subject comparison of effects of clear versus opaque bottles on maternal sensitivity and infant intake; order of bottle presentation was counterbalanced.
- Opaque Bottle Group - Clear Bottle Condition; Opaque Bottle Group - Opaque Bottle Condition: This group was given a set of opaque bottles to use during infant feedings for a full 12-week period. These mothers received everything provided to the clear group, but instead received 12 opaque bottles of various sizes (4-12 ounces). These bottles were stainless steel and compatible with a variety of different nipples manufactured by a leading bottle company. Mothers in the intervention group also received an additional handout that contained safety tips for their opaque bottles (e.g., never microwave your bottle).
  During post-tests, participants in both the Clear Bottle and Opaque Bottle Groups were asked to use the clear bottle during one feeding observation and the opaque bottle during the other feeding across the two post-test assessments, which ensured research assistants remained masked to whether the participant was in the intervention or control group and allowed for within-subject comparison of effects of clear versus opaque bottles on maternal sensitivity and infant intake; order of bottle presentation was counterbalanced.
Arm/Group | Clear Bottle Group - Clear Bottle Condition | Clear Bottle Group - Opaque Bottle Condition. | Opaque Bottle Group - Clear Bottle Condition | Opaque Bottle Group - Opaque Bottle Condition
Number analyzed (Participants) | 30 | 30 | 30 | 30
mL | 116.7 (10.1) | 119.5 (10.0) | 107.5 (10.2) | 114.9 (10.1)
Statistical Analysis 1: Comparison: Clear Bottle Group - Clear Bottle Condition vs Clear Bottle Group - Opaque Bottle Condition. vs Opaque Bottle Group - Clear Bottle Condition vs Opaque Bottle Group - Opaque Bottle Condition; Test type: Other — Repeated measures ANOVA was used to model between-subject effects of group (Clear versus Opaque), within-subjects effects of use of clear versus opaque bottles during the feeding observations, and potential group by bottle type interactions on infant intake during post-test feeding observations; p = 0.76, Mixed Models Analysis — Statistical significance was defined as p < 0.05; Models controlled for pre-test values, infant sex and age, time since last feeding, and whether the assessment was in-person or remote

2. Primary Outcome: Maternal Sensitivity to Infant Cues
Description: Mothers' behavior during feeding observations was coded using the Nursing Child Assessment Parent-Child Interaction - Feeding Scale (NCAFS). This scale contains six subscales, four of which describe maternal attributes (Sensitivity to Cues, Response to Child's Distress, Social-Emotional Growth Fostering, and Cognitive Growth Fostering) and two of which describe infant attributes (Clarity of Cues and Responsiveness to Caregiver). The present analysis focused on the Sensitivity to Cues subscale, which measures the degree to which the mother is able to understand and respond to her child's cues. This scale provides a global measure of how sensitive the mother is to the infant's needs during the feeding interaction. Possible score range is 0-16, which is derived from summing together maternal scores for each of the 16 subscale items. Higher scores indicate greater sensitivity to infant cues.
Time Frame: 12-week period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Clear Bottle Group - Clear Bottle Condition | Clear Bottle Group - Opaque Bottle Condition | Opaque Bottle Group - Clear Bottle Condition | Opaque Bottle Group - Opaque Bottle Condition
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale | 12.3 (0.4) | 12.6 (0.4) | 12.2 (0.4) | 12.2 (0.4)
Statistical Analysis 1: Comparison: Clear Bottle Group - Clear Bottle Condition vs Clear Bottle Group - Opaque Bottle Condition vs Opaque Bottle Group - Clear Bottle Condition vs Opaque Bottle Group - Opaque Bottle Condition; Test type: Other — Repeated measures ANOVA was used to model between-subject effects of group (Clear versus Opaque), within-subjects effects of use of clear versus opaque bottles during the feeding observations, and potential group by-bottle type interactions on maternal sensitivity during post-test feeding observations; p = 0.64, Mixed Models Analysis — Statistical significance was defined as p < 0.05; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Infant Weight-for-length Z-scores
Description: Infants' weight and length were assessed during home-based assessments. Infant weight and length were measured in triplicate using a portable infant scale/infantometer. To minimize bias, infants were always weighed and measured while only wearing a clean diaper and prior to the observed feeding.
  Weight and length values were standardized to age- and sex-specific weight-for-length z-scores based on the World Health Organization Child Growth Standards (https://www.who.int/tools/child-growth-standards). A z-score of 0 indicates that the child's weight status is at the population median; standard deviations closer to 0 represent healthier weight status. Standard deviations below 0 indicate the child's weight status is below the median, with values < -2 indicating the child is underweight. Standard deviations above 0 indicate the child's weight status is above the median, with values > 2 indicating the child is overweight or obese.
Time Frame: 12-week period
Population: Overall Number of Participants Analyzed for each group is not consistent with the number of participants indicated in the Participant Flow module because data were analyzed at the level of the dyad (n = 30 dyads per group), not at the level of each individual member of the dyad (n = 60 individuals per group, which represents 30 mothers + 30 infants). In addition, weight-for-length data were missing for n=12 dyads in the Clear Bottle Group and n=13 dyads in the Opaque Bottle Group.
Measure: Mean (Standard Error); unit: z-score
Groups:
- Clear Bottle Group: This group was given a set of clear bottles to use during infant feedings for a full 12-week period.These mothers received usual care from their pediatric providers and each mother was given 12 conventional, clear bottles of various sizes (4-12 ounces) that were compatible with a variety of different nipples manufactured by leading bottle companies. Mothers were also given handouts about proper formula preparation and paced bottle-feeding, which included messages about feeding in response to infant cues.
- Opaque Bottle Group: This group was given a set of opaque bottles to use during infant feedings for a full 12-week period. These mothers received everything provided to the clear group, but instead received 12 opaque bottles of various sizes (4-12 ounces). These bottles were stainless steel and compatible with a variety of different nipples manufactured by a leading bottle company. Mothers in the intervention group also received an additional handout that contained safety tips for their opaque bottles (e.g., never microwave your bottle).
Arm/Group | Clear Bottle Group | Opaque Bottle Group
Number analyzed (Participants) | 18 | 17
z-score | 0.22 (0.16) | 0.69 (0.15)
Statistical Analysis 1: Comparison: Clear Bottle Group vs Opaque Bottle Group; Test type: Other — General linear models were used to compare post-test weight-for-length z-scores (WLZ); p = 0.02, Regression, Linear — Statistical significance was defined as p < 0.05; These models controlled for baseline values (i.e., baseline WLZ), infant sex and age, and whether the assessment was in-person or remote

4. Secondary Outcome: Change in Infant Waist Circumference
Description: Infant central adiposity was assessed via a waist circumference measurement, which was assessed during home-based assessments by trained research assistants. Waist circumference was assessed in triplicate using a study-specific Gulick II tape measure.
Time Frame: 12-week period
Population: Overall Number of Participants Analyzed for each group is not consistent with the number of participants indicated in the Participant Flow module because data were analyzed at the level of the dyad (n = 30 dyads per group), not at the level of each individual member of the dyad (n = 60 individuals per group, which represents 30 mothers + 30 infants). In addition, waist circumference data could not be obtained for n=16 dyads in the Clear Bottle Group and n=16 dyads in the Opaque Bottle Group.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Groups:
- Clear Bottle Group: This group was given a set of clear bottles to use during infant feedings for a full 12-week period. These mothers received usual care from their pediatric providers and each mother was given 12 conventional, clear bottles of various sizes (4-12 ounces) that were compatible with a variety of different nipples manufactured by leading bottle companies. Mothers were also given handouts about proper formula preparation and paced bottle-feeding, which included messages about feeding in response to infant cues.
Arm/Group | Clear Bottle Group | Opaque Bottle Group
Number analyzed (Participants) | 14 | 14
centimeters | 44.7 (0.59) | 43.1 (0.63)
Statistical Analysis 1: Comparison: Clear Bottle Group vs Opaque Bottle Group; Test type: Other — General linear models were used to compare post-test waist circumference for the Clear versus Opaque groups; p = 0.07, Regression, Linear — Statistical significance was defined as p < 0.05; Model controlled for baseline values (i.e., waist circumference), infant sex and age, and whether the assessment was in-person or remote

5. Secondary Outcome: Change in Infant Triceps Skinfolds z-Scores
Description: Triceps skinfold thickness, a marker of infant adiposity, was assessed during home-based assessments by trained research assistants. A study-specific Harpenden caliper was used for this assessment.
  Triceps skinfold thickness values were standardized to age- and sex-specific z-scores based on the World Health Organization Child Growth Standards (https://www.who.int/tools/child-growth-standards). A z-score of 0 indicates that the child's adiposity is at the population median. Standard deviations below 0 indicate the child's adiposity is below the median and standard deviations above 0 indicate the child's adiposity is above the median. Standard deviations closer to 0 represent healthier levels of adiposity.
Time Frame: 12-week period
Population: Overall Number of Participants Analyzed for each group is not consistent with the number of participants indicated in the Participant Flow module because data were analyzed at the level of the dyad (n = 30 dyads per group), not at the level of each individual member of the dyad (n = 60 individuals per group, which represents 30 mothers + 30 infants). In addition, skinfold data could not be obtained for n=23 dyads in the Clear Bottle Group and n=23 dyads in the Opaque Bottle Group.
Measure: Least Squares Mean (Standard Error); unit: z-scores
Arm/Group | Clear Bottle Group | Opaque Bottle Group
Number analyzed (Participants) | 7 | 7
z-scores | -0.52 (0.40) | -0.77 (0.47)
Statistical Analysis 1: Comparison: Clear Bottle Group vs Opaque Bottle Group; Test type: Other — General linear models were used to compare post-test triceps skinfold z-scores for the Clear versus Opaque groups; p = 0.70, Regression, Linear — Statistical significance was defined as p < 0.05; Model controlled for baseline values (i.e.,triceps skinfolds z-scores), infant sex and age, and whether the assessment was in-person or remote

6. Secondary Outcome: Change in Infant Subscapular Skinfolds z-Scores
Description: Subscapular skinfold thickness, a marker of infant adiposity, was assessed during home-based assessments by trained research assistants. A study-specific Harpenden caliper was used for this assessment.
  Subscapular skinfold thickness values were standardized to age- and sex-specific z-scores based on the World Health Organization Child Growth Standards (https://www.who.int/tools/child-growth-standards). A z-score of 0 indicates that the child's adiposity is at the population median. Standard deviations below 0 indicate the child's adiposity is below the median and standard deviations above 0 indicate the child's adiposity is above the median. Standard deviations closer to 0 represent healthier levels of adiposity.
Time Frame: 12-week period
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: z-scores
Arm/Group | Clear Bottle Group | Opaque Bottle Group
Number analyzed (Participants) | 7 | 7
z-scores | 0.67 (0.22) | 0.37 (0.25)

7. Secondary Outcome: Mothers' Perceptions of the Bottles
Description: Mothers' perceptions of their assigned bottles, including any perceived barriers to their use, were assessed via a questionnaire developed by the investigators.
Time Frame: 12-week period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Bottle Group | Opaque Bottle Group
Number analyzed (Participants) | 30 | 30
Participants
  indicated they would continue to use their assigned bottle after the study ended | 24 | 24
  indicated they would not continue to use their assigned bottle after the study ended | 6 | 6

ADVERSE EVENTS:
Time Frame: 3-5 months after randomization
Description: Definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definitions.
Groups:
- Clear Bottle Group - Mothers; Clear Bottle Group - Infants: This group was given a set of clear bottles to use during infant feedings for a full 12-week period. These mothers received usual care from their pediatric providers and each mother was given 12 conventional, clear bottles of various sizes (4-12 ounces) that were compatible with a variety of different nipples manufactured by leading bottle companies. Mothers were also given handouts about proper formula preparation and paced bottle-feeding, which included messages about feeding in response to infant cues.
- Opaque Bottle Group - Mothers; Opaque Bottle Group - Infants: This group was given a set of opaque bottles to use during infant feedings for a full 12-week period. These mothers received everything provided to the clear group, but instead received 12 opaque bottles of various sizes (4-12 ounces). These bottles were stainless steel and compatible with a variety of different nipples manufactured by a leading bottle company. Mothers in the intervention group also received an additional handout that contained safety tips for their opaque bottles (e.g., never microwave your bottle).
Arm/Group | Clear Bottle Group - Mothers | Clear Bottle Group - Infants | Opaque Bottle Group - Mothers | Opaque Bottle Group - Infants
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/38

LIMITATIONS AND CAVEATS:
This study consisted of mothers who were exclusively or predominantly bottle-feeding. We were unable to obtain an objective assessment of adherence, daily feeding patterns, or detailed information regarding the extent to which non-maternal caregivers (e.g., fathers, daycare providers) used clear versus opaque bottles with infants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03711370/Prot_SAP_ICF_000.pdf